CLINICAL TRIAL: NCT02979041
Title: Therapeutic Virtual Reality Training for Neck Pain in Israeli Air Force Pilots - A Randomized Controlled Trial
Brief Title: VR Training for Pilots With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Medical Corps, Israel Defense Force (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHaifaAF
Record Dates: First submitted 2016-10-05; First posted 2016-12-01 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2016-06

CONDITIONS: Neck Pain; Cervical Pain
Keywords: neck pain; Virtual reality; Range of motion; physiotherapy; Air force; kinematics
MeSH Terms: conditions — Neck Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Active Comparator): Patients in the control group will receive standard physiotherapy and medical care, as provided to all patients with neck pain in the aviation medicine clinic. This will reflect the standard care that has been provided to all patients.
  Interventions: Other: Standard Care
- intervention (Experimental): Standard care (as provided to controls) with the addition of virtual reality training (a self-exercise program) using a VR system to address the fast, accurate head control required in flying tasks.
  Interventions: Behavioral: Interactive virtual reality training

INTERVENTIONS:
Behavioral: Interactive virtual reality training — The proposed VR intervention program will provide active training to be performed individually 4 times a week for 20 minutes a session.
  The intervention program will be supervised by qualified, experienced physiotherapists, and will include individual training and two follow up meetings during the study period. The intervention program will include strengthening and endurance exercises for the cervical and shoulder girdle muscles. Training will include sensorimotor control and functional, quick, accurate, neck motion, using interactive VR training systems. This type of advanced training is very relevant to the pilots function in the cockpit as it includes interactive tasks aimed to increase range, speed, smoothness, accuracy, and control of cervical motion.
  Arms: intervention
Other: Standard Care — physiotherapy and medical care as provided currently
  Arms: control

SUMMARY:
The aim of the proposed study is to investigate the effectiveness of an interactive, virtual reality (VR) training program for pilots compared with standard care. The study will be a randomized controlled trial (RCT) consisting of 60 pilots randomized into one of two groups: standard physiotherapy and medical care vs standard care and VR training. Outcome measures will include subjective scores of pain intensity and global perceived effect; objective measures of range of motion (ROM), neck motion velocity, and motion accuracy; and functional measure of days grounded due to neck pain. Data will be analyzed using ANOVA for within and between groups analyses.

DETAILED DESCRIPTION:
The aim of the proposed study is to investigate the effectiveness of an interactive, virtual reality (VR) training program for pilots compared with standard care. The proposed intervention program includes training in neck range of motion, control, accuracy and coordination and is expected to reduce the prevalence and operational impact of neck pain in the intervention group more effectively than does standard care alone.

The proposed study will be designed as a randomized, controlled trial (RCT). Sixty fighter and helicopter pilots will be randomized into two groups, to receive either standard physiotherapy and medical care or standard care with the addition of interactive, dynamic, controlled training (a self-exercise program) in VR to address the fast, accurate head control required in flying tasks.

Subjective outcome measures will include pain intensity and global perceived effect. Objective measures will include range of motion, motion velocity and accuracy. The functional measure will include days grounded due to neck pain.

Statistical analysis will use independent, repeated measures ANOVA on each parameter, within and between groups. Post hoc comparisons, including several preplanned contrasts, will be performed to assess differences before and after treatment, and the stability of changes over time, in each group. The relationship of risk factors to performance failures will be assessed using multivariate logistic regression analyses.

This study is the first in the Israeli Air Force to evaluate this type of comprehensive, functional intervention program. Such research will dramatically advance the military's health care approach to neck pain, and may be further applied to other populations in and outside the Israeli Defence Force (IDF). This study may serve as a stepping stone to further research related to diagnosis, treatment, and prevention methods during a pilot's active service.

ELIGIBILITY:
Inclusion Criteria:

* fighter and helicopter pilots from the Israeli Air Force
* acute, sub-acute, and chronic neck pain, with or without referral to the upper limbs

Exclusion Criteria:

* neurological disorders (e.g. evidence for positive neurological signs), systemic disease, history of spinal surgery, or any disorders that may limit the ability to exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-09-01; Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity is measured using the Visual Analogue Scale (VAS, 0-100mm) | change from baseline at 4 weeks, 3 and 6 months.
  Pain intensity was measured using the Visual Analogue Scale (VAS, 0-100mm)
Global perceived effect of the provided treatment is measured on a scale from -5 to +5. | change from baseline at 4 weeks, 3 and 6 months.
  Global perceived effect of the provided treatment was measured on a scale from -5 to +5. Zero represented no change, +5 excellent improvement due to the treatment provided, and -5, vast worsening.
Functional outcome is measured by the number of grounding days from flying due to neck pain. | change from baseline at 4 weeks, 3 and 6 months.
  The number of days the pilot was grounded due to neck pain.

SECONDARY OUTCOMES:
Cervical range of motion is measured using the neck VR system (ROM, degrees) | change from baseline at 4 weeks, 3 and 6 months.
  Cervical range of motion (ROM, degrees) is measured using the neck VR system, into flexion, extension, right and left rotation.
Cervical motion velocity is measured using the neck VR system (degrees/second) | change from baseline at 4 weeks, 3 and 6 months.
  Cervical motion velocity is measured using the neck VR system (degrees/second) into flexion, extension, right and left rotation.
Cervical muscles isometric strength is measures using a dynamometer (Newton) | change from baseline at 4 weeks, 3 and 6 months.
  Cervical muscles isometric strength is measures using a dynamometer (Newton), in the directions of static flexion and extension.

CONTACTS AND LOCATIONS:
Overall Officials: Hilla Sarig-Bahat, PT, PhD, Principal Investigator — Department of Physical Therapy, University of Haifa
Locations (2):
- Israel (2):
  - The Faculty of Social Welfare and Health Sciences, Haifa
  - Medical Aviation Unit, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van den Oord MH, De Loose V, Meeuwsen T, Sluiter JK, Frings-Dresen MH. Neck pain in military helicopter pilots: prevalence and associated factors. Mil Med. 2010 Jan;175(1):55-60. doi: 10.7205/milmed-d-09-00038. PMID 20108843
- [Background] Tucker B, Netto K, Hampson G, Oppermann B, Aisbett B. Predicting neck pain in Royal Australian Air Force fighter pilots. Mil Med. 2012 Apr;177(4):444-50. doi: 10.7205/milmed-d-11-00256. PMID 22594136
- [Background] Grossman A, Nakdimon I, Chapnik L, Levy Y. Back symptoms in aviators flying different aircraft. Aviat Space Environ Med. 2012 Jul;83(7):702-5. doi: 10.3357/asem.3225.2012. PMID 22779315
- [Background] Knudson R, McMillan D, Doucette D, Seidel M. A comparative study of G-induced neck injury in pilots of the F/A-18, A-7, and A-4. Aviat Space Environ Med. 1988 Aug;59(8):758-60. PMID 3178626
- [Background] Sarig Bahat H, Weiss PL, Laufer Y. The effect of neck pain on cervical kinematics, as assessed in a virtual environment. Arch Phys Med Rehabil. 2010 Dec;91(12):1884-90. doi: 10.1016/j.apmr.2010.09.007. PMID 21112430
- [Background] Jones JA, Hart SF, Baskin DS, Effenhauser R, Johnson SL, Novas MA, Jennings R, Davis J. Human and behavioral factors contributing to spine-based neurological cockpit injuries in pilots of high-performance aircraft: recommendations for management and prevention. Mil Med. 2000 Jan;165(1):6-12. PMID 10658420
- [Background] Ang BO, Monnier A, Harms-Ringdahl K. Neck/shoulder exercise for neck pain in air force helicopter pilots: a randomized controlled trial. Spine (Phila Pa 1976). 2009 Jul 15;34(16):E544-51. doi: 10.1097/BRS.0b013e3181aa6870. PMID 19770596
- [Background] Alricsson M, Harms-Ringdahl K, Larsson B, Linder J, Werner S. Neck muscle strength and endurance in fighter pilots: effects of a supervised training program. Aviat Space Environ Med. 2004 Jan;75(1):23-8. PMID 14736129
- [Background] Hamalainen O, Heinijoki H, Vanharanta H. Neck training and +Gz-related neck pain: a preliminary study. Mil Med. 1998 Oct;163(10):707-8. PMID 9795549
- [Background] Sarig Bahat H, Takasaki H, Chen X, Bet-Or Y, Treleaven J. Cervical kinematic training with and without interactive VR training for chronic neck pain - a randomized clinical trial. Man Ther. 2015 Feb;20(1):68-78. doi: 10.1016/j.math.2014.06.008. Epub 2014 Jul 5. PMID 25066503